CLINICAL TRIAL: NCT02393573
Title: Attenuating The Post-Operative Insulin Resistance And Promoting Protein Anabolism In Patients Undergoing Major Lung or Abdominal Surgery
Brief Title: Attenuating The Post-Operative Insulin Resistance And Promoting Protein Anabolism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Mitacs (Industry); Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Dr. Liane S. Feldman, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-264-SDR
Record Dates: First submitted 2015-02-10; First posted 2015-03-19 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Pre-Diabetes; Major Lung or Abdominal Surgery; Insulin Resistance
Keywords: Insulin Resistance; Protein balance; Surgery; Post operative complications; metformin; Pre-diabetes; Fasting blood glucose
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): Metformin will be administered as pills to be taken orally with an initial dose of 850 mg on the first day; the dose will be increased to 850 mg every 12 hours and 850mg every 8 hours respectively on the second day and then on the days to follow up to the morning of the surgery. Metformin will be discontinued on the day of surgery and will be restarted immediately after surgery.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo will be administered exactly in the similar way to Metformin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Patients will take metformin for two weeks before Surgery and 2 days after the surgery
  Arms: Metformin
Drug: Placebo — Patients will take Placebo pills for two weeks before Surgery and 2 days after the surgery
  Arms: Placebo

SUMMARY:
Major surgery results in a stress- induced catabolic response, marked by post-operative insulin resistance, hyperglycemia and loss of body protein, which is associated with increased morbidity, mortality and adverse outcomes. There has been a great deal of research on different approaches to optimize post-operative insulin sensitivity including hormonal and nutritional interventions, minimally invasive surgical techniques and epidural anesthesia. However, the correlation between insulin resistance and body protein loss is not well understood. Metformin is the most widely used insulin sensitizing and blood glucose-lowering drug in treatment of type 2 diabetic patients. This study will: 1) estimate the correlation between insulin resistance and body protein loss in pre-diabetic lung/colorectal resection patients; 2) investigate whether the post-operative metabolic state can be improved by the pre-operative administration of metformin; and assess the impact of metformin on surgical complications and hospital length of stay. The results of this study will provide insight into the relationship between insulin resistance and post-operative adverse events and potentially suggest a novel approach to improve outcomes using Metformin, a drug already in wide clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Elective open anatomic lung resections: segmentectomy, lobectomy, bi-lobectomy
2. Colorectal surgery for non-metastatic disease (including right, transverse, left, sigmoid, subtotal, total, and hemicolectomy)
3. Primary or secondary lung cancer
4. At least 18 years of age with
5. HbA1c 5.7- 6.5 %
6. Not receiving any kind of glucose lowering medication.

Exclusion Criteria:

1. Already diagnosed with diabetes (Hb A1c > 6.5%)
2. Are pre-diabetic receiving glucose lowering intervention ( any glucose lowering medication)
3. Have renal or liver dysfunction (serum creatinine above 124 micromol/L in women and 133 micromol/L in men, bilirubin >50 micromol/L)
4. will undergo extended resection of adjacent organs, chest wall resections, bronchoplasty, non-anatomic lung resections
5. Will undergo Pneumonectomy
6. Non-elective operations
7. Have mental conditions (e.g. dementia, disabling orthopedic and neuromuscular disease, psychosis),
8. Have cardiac abnormalities, severe end-organ disease such as cardiac failure (New York Heart Association classes III-IV), Chronic obstructive pulmonary disease(COPD), sepsis, morbid obesity (BMI >40 kg/m2), anemia (hematocrit < 30 %, hemoglobin <100g/L albumin < 25mg/dl)
9. Have received steroids for longer than 30 days
10. Have poor English or French comprehension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-11; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in fasting blood glucose | 2 weeks before surgery (pre-operative) and on the morning before the surgery and every morning after the surgery (post operative) for three days or until discharge which ever comes earlier
  the level of plasma glucose after 6 hours of fasting

SECONDARY OUTCOMES:
Change in whole body protein balance | 2 weeks before surgery (pre-operative) and hours after the surgery (post operative)
  The difference between the Pre-operative whole body protein balance( prior to metformin treatment) and the post operative whole body protein balance
Comparing the Homeostasis model assessment (HOMA) index at three different time points ( by employing Fasting blood sugar and Plasma Insulin) | at 3 time points as follow : 2 weeks before surgery, on the day of surgery and 48 hours after the surgery
glycosylated Hba1c | 2 weeks before surgery
  plasma level of glycosylated Hba1c
Comparing the pre-operative body impedance and the post operative body impedance (to asses the body composition specifically the amount of body fat) | 2 weeks before surgery and 48 hours after the surgery
  Measures body composition specifically fat content
Surgical Complications | 30 days after operation
  Any complication related to the surgery with in 30 days post operation
length of hospital stay | Up to 30 days after operation
  Length of hospital stay is calculated as the total length of hospitalization from the date of admission for the purpose of surgery until the date of discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Liane Feldman, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Francesco Carli, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada